CLINICAL TRIAL: NCT07208162
Title: Adapting the SHARE for Dementia Early-Stage Dyadic Intervention: A Stage I Pilot Study With African-American Families
Brief Title: SHARE Adaptation Intervention for African-American Families
Acronym: SHARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benjamin Rose Institute on Aging (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRIA2025SHARE-ROYBAL; 1P30AG086562-01 (NIH)
Record Dates: First submitted 2025-08-21; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Mild Dementia; Moderate Dementia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two groups: Treatment (SHARE) and Control (Treatment as usual single session)
Masking Description: Research interviewers will be blinded to condition at Baseline (Time 1) only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (SHARE Dyadic Intervention) (Experimental): Treatment group dyads are comprised of a PLWD with mild to moderate dementia and his/her preferred CG. Following recruitment and the consent process and screening, baseline telephone interviews (T1) with trained interviewers from the Benjamin Rose Institute on Aging will be completed separately with all CGs and PLWDs. Treatment group dyads will receive the culturally adapted SHARE intervention compromised of up to five, 60- 90-minute, curriculum-guided sessions with a SHARE Counselor over a 8-10 week period. A (T2) follow-up interview will be conducted approximately two weeks after treatment group dyads complete their final session;.
  Interventions: Behavioral: 5+1 Adapted, early-stage dyadic care planning intervention
- Control (Treatment as usual single session) (Active Comparator): Control group dyads are comprised of a PLWD with mild to moderate dementia and his/her preferred CG. Following recruitment and the consent process and screening, baseline telephone interviews (T1) with trained interviewers from the Benjamin Rose Institute on Aging will be completed separately with all CGs and PLWDs. Control group participants will receive a treatment as usual equivalent: a standardized educational and resource single session with a packet of information. A (T2) follow-up interview will be conducted approximately approximately eight weeks after (T1) baseline interviews.
  Interventions: Behavioral: Counseling session and printed resources

INTERVENTIONS:
Behavioral: 5+1 Adapted, early-stage dyadic care planning intervention — The intervention group will receive the adapted SHARE Dyadic program, consisting of five, 60-90-minute curriculum-guided sessions with a SHARE Counselor, plus one optional family session.
  Arms: Treatment (SHARE Dyadic Intervention)
Behavioral: Counseling session and printed resources — Control group participants will receive a treatment as usual equivalent: a single, standardized educational and resource session with a packet of information.
  Arms: Control (Treatment as usual single session)

SUMMARY:
This project aims to culturally adapt the SHARE program for African-Americans in early-moderate stage dementia and their care partner. Upon completion of the adaptation, a pilot randomized-control trial wil be confucted to compare the adaptaed SHARE program versus usual care.

DETAILED DESCRIPTION:
Aim 1: Review SHARE for Dementia materials with an Advisory Committee (AC; 6-10 African Americans with lived experience and experts) to identify distinct needs of African American care dyads and culturally adapt SHARE using this input. Deliverables: Develop SHARE V1 Culturally tailored V1 SHARE Counselor Manual, V1 SHARE Guide for Families, and V1 SHARE Counselor training Aim 2: Conduct focus groups with African American care dyads (n=2 groups; n=10 dyads total, or until saturation) and community service provider staff (n= 2 groups; n=10, or until saturation) to identify strengths and limitations of the V1 SHARE materials, procedures, and protocols. Deliverables: SHARE for African Americans (Version 2;V2); Culturally tailored V2 SHARE Counselor Manual, V2 SHARE Guide for Families, and V2 SHARE Counselor training Aim 3: Train SHARE counselors (n=20) to implement V2 of SHARE. Aim 4: Examine: a) the acceptability and feasibility and; 2) preliminary efficacy of the culturally adapted V2 of SHARE in a fully powered trial with 120 African American care dyads.

ELIGIBILITY:
Inclusion Criteria:

* African American dyads (both the caregivers and the care-recipient, an individual with an early-stage memory impairing condition (e.g., Alzheimer's disease, vascular dementia, cognitive impairment, etc.)
* Care-recipient lives at home.
* The caregiver (CG) and/or the person with dementia (PWD), or symptoms of memory loss must identify as African American.
* PWD must be at least 50 years old and CGs 18 or older,
* Ability to speak and read English,
* Experiencing signs and symptoms of mild to moderate dementia through family caregiver report on the Dementia Severity Rating Scale and meeting the National Institute on Aging and the Alzheimer's Association clinical criteria for probable AD.

Exclusion Criteria:

* A mental health condition (e.g., schizophrenia, bipolar disorder, major depression)
* A traumatic brain injury
* Intellectual or developmental disability
* Individuals experiencing extreme difficulty adjusting and coping to the diagnosis • Individuals living in an institutional setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Session length | After each session; within 10 weeks of baseline.
  SHARE counselors will report length of each session, and we will determine the number of sessions conducted were within 60-90 minutes - the prescribed treatment protocol.
Attendance | After each session; within 10 weeks of baseline.
  SHARE counselors will report the number of sessions attended out of 6 treatment sessions offered.
Attrition | Follow up (T2); within 12 weeks of baseline.
  We will assess the number of caregivers and PLWD retained at follow-up
Satisfaction with session | After each session; within 10 weeks of baseline.
  Caregivers and PLWD will be asked about their satisfaction with SHARE regarding the: 1) experience; 2) counselor; 3) materials; 4) sessions; 5) postintervention relationship functioning.
Treatment process | Follow up (T2); within 12-weeks of baseline.
  Caregivers and PLWD will be asked to agree or disagree with statements about SHARE Counselor, understanding of choices, knowledge of dementia, connection to care partner.
Overall satisfaction | Follow up (T2); within 12 weeks of baseline.
  Caregivers and PLWD will be asked to rate their satisfaction with care values and preferences discussions, spacing between sessions, importance of knowledge gained, etc.
Utility | Follow up (T2); within 12 weeks of baseline.
  Caregivers and PLWD will be asked to rate the usefulness of materials and information shared, skill of counselor, commitment to care plan.
Feasibility of SHARE | Follow up (T2); within 12 weeks of baseline.
  Caregivers and PLWD will be asked about the appropriateness of time spent in session and number of sessions.
Acceptability | Follow up (T2); within 12 weeks of baseline.
  Caregivers and PLWD will be asked about the main benefits and drawbacks of SHARE.
Goals | Follow up (T2); within 12 weeks of baseline.
  Caregivers and PLWD will be asked to indicate their goals of participating in SHARE, such as: Dementia education, communication skills, knowledge of resources, building a network of support, etc.

SECONDARY OUTCOMES:
Dyadic Relationship Scale (DRS) (Clinical Outcomes (Distal Effects; Secondary)) | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  The Dyadic Relationship Scale consists of 28 items that asks care partners and PLWD how often of the time (15-items), and how often in the past month (13-items), they think a statement applies to their relationship. Responses are (0-3) ranging from "All or nearly all of the time" to "None or almost none of the time". Ranges are a total of 0-84, with higher scores indicating more positive dyadic relationship.
Personal and Instrumental Activities of Daily Living (PIADL) | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  The Personal and Instrument Activities of Daily Living is a an 18-item measure that asks care partners to rate the PLWD ability to perform daily activities. Responses are (1) Does by self/ Needs no help, (2) Needs reminders/ Needs a little help, (3) Needs help most of the time, and (4) Needs help all the time (unable to do activity). Range is from 18-72, with lower scores indicating less ability of PLWD to perform daily activities independently.
Emotional-Intimacy Disruptive Behavior Scale (EIDBS) | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  The Emotional-Intimacy Disruptive Behavior Scale is a an 8-item measure to asks care givers and PLWD to assess the extent care partners with hold or distort symptoms or feelings to protect their care partner. Response options are (1) None of the time, (2) Some of the time, (3) Much of the time, (4) Most or all of the time. Range is from 8-32, with higher scores indicating higher distortions of feelings
Dementia Quality of Life +/- Affect | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  Caregivers and PLWD will be asked six positive/six negative affect indicators.
Center for Epidemiological Studies Depression Scale (CES-D) | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  Caregivers and PLWD will be asked to respond to a 20-item measure of how often in past week they experience depressive symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Stress in Providing Care | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  Caregivers will be asked open-ended questions.
Leisure & Healthy Behaviors | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  Caregivers and PLWD will complete an inventory of enjoyable activities and self-care practices.
Quality of Life - AD (QoL-AD) | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  Caregivers and PLWD will respond to a 13-item questionnaire designed to provide a report of the quality of life for the PLWD participant. Response options are from 1 (Poor) - (4) excellent for each item. Range from 13-52, higher scores indicate higher quality of life.

OTHER OUTCOMES:
Self-Care education (Mechanisms (Proximal Effects; Secondary)) | After each session; within 10 weeks of baseline.
  SHARE counselors will report on dyad's self-care strengths and challenges after sessions 1 & 4 of the treatment intervention.
Communication skills (Mechanisms (Proximal Effects; Secondary)) | After each session; within 10 weeks of baseline.
  Communication skills are 4-items that counselors respond to after each session of the treatment intervention to rate the degree of which care partner and PLWD communicated with the counselor, as well as to rate the quality and balance of amount of talking that occurred during the sessions. Response options range from 1 "Not at all" to 7 "very", with higher scores indicating better communication.
Knowledge of Available Service; Service Availability Measure (Mechanisms (Proximal Effects; Secondary)) | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  The Knowledge of Available Service subscale of the Service Availability Measure is a 14-item measure of the PLWD and their care partner's knowledge of different community of mental health services available. Response are (1) yes and (0) no. Range is 0-14, with higher scores indicating higher knowledge of services available.
Use of Services; Service Availability Measure (Mechanisms (Proximal Effects; Secondary)) | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  The Use of Services subscale of the Service Availability Measure is a 14-item measure of the PLWD and their care partner's use of different community of mental health services available in the past 3 months. Response are (1) yes and (0) no. Range is 0-14, with higher scores indicating higher use of services available.
Care Values; Care Values Scale (CVS) (Mechanisms (Proximal Effects; Secondary)) | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  The Care Values Scale is a 25-item measure to capture what the PLWD, and their care partners, think are most important to the PLWD's future care. Response options are (1) Not at all important, (2) Somewhat important, (3) Very important. Range is 25-75, with higher scores indicating higher levels of importance to the various domains of care asked.
Preferences for Care Tasks; Preferences for Care Tasks Scale (PCTS) (Mechanisms (Proximal Effects; Secondary)) | Baseline (T1), Follow up (T2); within 12 weeks of baseline.
  The Preferences for Care Tasks Scale is a 19-item measure to capture who the PLWD, and their care partners believe the PLWD, prefers to help them with various care tasks. Response options are (1) the care giver, (2) friends or other family, (3) paid professional help. Range is 19-57, with higher scores indicating higher preferences that care tasks are performed outside of the dyad.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Orsulic-Jeras, Principal Investigator — Benjamin Rose Institute on Aging
Locations (1):
- Benjamin Rose, Cleveland, Ohio, United States

DOCUMENTS (2):
  • Study Protocol (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT07208162/Prot_000.pdf
  • Informed Consent Form (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT07208162/ICF_001.pdf